CLINICAL TRIAL: NCT07365891
Title: Help-Seeking Behavior in Cases of Emotional Neglect: The Decision-Making Process of Adolescents in Dutch-Speaking Secondary Education in Brussels
Brief Title: Recognizing Emotional Neglect and Help-Seeking Intention Among Adolescents in Brussels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Fiona Roulent, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25276_Hulpzoekgedrag
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adolescents in School-based Population; Emotional Neglect; Help-Seeking Behavior
Keywords: Help-seeking; Decision-making; Emotional neglect; Adolescents; Secondary education; Recognition; Help-seeking behavior; Child neglect; Child maltreatment and neglect
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Interventional study employing vignettes to examine adolescents' recognition of emotional neglect and help-seeking behavior
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- boy x clear situation (Experimental): Participants are exposed to a vignette describing a boy in a clear emotional neglect situation.
  Interventions: Behavioral: Emotional neglect vignettes
- boy x ambiguous situation (Experimental): Participants are exposed to a vignette describing a boy in a ambiguous emotional neglect situation.
  Interventions: Behavioral: Emotional neglect vignettes
- girl x ambiguous situation (Experimental): Participants are exposed to a vignette describing a girl in a ambiguous emotional neglect situation.
  Interventions: Behavioral: Emotional neglect vignettes
- girl x clear situation (Experimental): Participants are exposed to a vignette describing a girl in a clear emotional neglect situation.
  Interventions: Behavioral: Emotional neglect vignettes

INTERVENTIONS:
Behavioral: Emotional neglect vignettes — Participants are randomly assigned to one of four written vignettes of adolescents experiencing emotional neglect. Each vignette differs by gender (boy or girl) and by situation clarity (ambiguous or clear).

SUMMARY:
The goal of this study is to find out how well adolescents in Dutch-speaking secondary schools in Brussels can recognize emotional neglect, and how this relates to their intention to seek help.

The main research questions are:

1. How well do adolescents recognize situations of emotional neglect, and do boys and girls differ in their recognition?
2. Does recognition of emotional neglect predict adolescents' intention to seek help?

This study is conducted through an online survey. Participants will read one of four short written stories about an adolescent experiencing emotional neglect. The stories vary by gender (boy or girl) and by the clarity of the neglect (clear or ambiguous). After reading, participants answer questions about the story, including their thoughts and how they might respond in a similar situation. They also answer questions about their own experiences and attitudes toward help-seeking.

ELIGIBILITY:
Inclusion Criteria:

* Age: adolescents aged 11-25 years;
* Education: enrolled in regular full-time secondary education;
* School location: Brussels-Capital Region;
* School language: Dutch;
* Consent: informed consent provided by the adolescent and their parent(s)/guardian.

Exclusion Criteria:

* Age: younger than 11 years or older than 25 years;
* Education: not enrolled in regular full-time secondary education;
* School location: outside the Brussels-Capital Region;
* School language: non - Dutch-speaking;
* Consent: informed consent not provided by the adolescent or their parent(s)/guardian.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recognition of emotional neglect | Immediately after reading the vignette
  Recognition is measured by asking participants to indicate whether emotional neglect is present in the vignette, using a 4-point Likert scale (1 = definitely not, 2 = probably not, 3 = probably yes, 4 = definitely yes). Higher scores indicate greater recognition of emotional neglect.
  Scores will be analyzed using analysis of covariance (ANCOVA) with age as a covariate. Factors include participant gender (boy or girl), vignette gender (boy or girl), and type of situation (ambiguous or clear).
  Exploratory analyses may examine recognition of other types of maltreatment (physical abuse, physical neglect, emotional abuse, and sexual abuse).
Help-seeking intention | Immediately after reading the vignette
  Help-seeking intention is measured by asking participants to indicate whether they would seek help in the situation described in the vignette, using a 4-point Likert scale (1 = definitely not, 2 = probably not, 3 = probably yes, 4 = definitely yes). Higher scores indicate greater intention to seek help.
  Scores will be analyzed using linear regression, with recognition as the independent variable and help-seeking intention as the dependent variable. Additional analyses will test whether perceived severity and anticipated risk of future harm moderate the relationship between recognition and help-seeking intention.

SECONDARY OUTCOMES:
Severity | Immediately after reading the vignette
  Severity is measured by asking participants to indicate how severe they perceived the situation described in the vignette, using a 4-point Likert scale (1 = not at all severe, 2 = not severe, 3 = severe, 4 = very severe). Higher scores indicate greater perceived severity.
Risk of future harm | Immediately after reading the vignette
  Risk of future harm is measured by asking participants to estimate the probability that the adolescent in the vignette will experience future physical or emotional problems. Each type of problem is rated on a 6-point Likert scale (1 = no chance, 2 = very small chance, 3 = small chance, 4 = moderate chance, 5 = large chance, 6 = very large chance). Higher scores indicate greater anticipated risk of future harm.

IPD SHARING:
Plan to Share IPD: No